CLINICAL TRIAL: NCT00749814
Title: Sleep Disturbances in Hospitalized Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Yakov Sivan, Tel Aviv Sourasky Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-08-YS-371-CTIL
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-08

CONDITIONS: Sleep Disorders
Keywords: sleep patterns in children in the night prior to surgery and post surgery.; the influence of melatonin on sleep patterns
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- A (Experimental): Study group will receive melatonin.
  Interventions: Dietary Supplement: Melatonin
- B (Placebo Comparator): Placebo
  Interventions: Other: Placebo tablets
- C (No Intervention): No intervention control group.

INTERVENTIONS:
Dietary Supplement: Melatonin — Melatonin slow release tablets, 2 mg, 1 hour before bedtime for 7 days prior to admission to the hospital and up to 7 days after surgery.
  Other Names: Circadin (melatonin 2 mg)
  Arms: A
Other: Placebo tablets — Placebo
  Arms: B

SUMMARY:
Background

Sleep disturbances are prevalent in hospitalized adult patients manifested as reduced sleep time and sleep efficiency as well as increased awakenings. Insomnia is the most frequent sleep disturbance. The effect of the change in sleep patterns in children prior to and after an elective surgery has not been evaluated objectively. Sleep in hospital may influence biological processes related to circadian rhythm.

Melatonin is a hormone secreted by the pineal gland in a diurnal rhythm regulated by light- light suppresses melatonin secretion, while darkness enhances it. Melatonin has both chrono-biotic and sleep promoting properties. Exogenous administration of melatonin shortens sleep latency, increases sleep efficiency and total sleep time. Melatonin also improves disrupted circadian rhythm. Melatonin promotes sleep in a similar way to the natural sleep process, and maintains normal sleep architecture.

Melatonin has a positive effect on children with sleep disturbances and is routinely administrated in pediatric sleep centers around the world for insomnia and a variety of sleep disorders. Side effects of melatonin are rare and scarce. Circadin is a slow released formulation of melatonin, which mimics night time secretion of natural melatonin. Children with sleep disorders who were treated with controlled release melatonin, demonstrated improvement in sleep latency and total sleep time.

It is reasonable to assume that hospitalized children have disturbed sleep patterns prior to and following elective surgery. We hypothesize that melatonin will improve sleep patterns prior to and following surgery, by reducing sleep latency and extending total sleep time. We also hypothesize that this improvement will have positive impact on anesthetic stress measures and on recovery.

The purposes of the study are: 1. To characterize sleep patterns in children undergoing surgery on the admission night prior to surgery; 2. To evaluate the effect of melatonin on sleep parameters on the night prior to surgery in children; 3. To evaluate the effect of melatonin on physiologic stress parameters during anesthesia and surgery in children; 4. To evaluate the effect of melatonin on sleep parameters of children postoperatively; 5. To evaluate the effect of melatonin on postoperative outcome measures in children.

Patients, Methods. Ninety children (aged 4-18 years) will be evaluated. Sleep disorders will be screened by a pediatric sleep questionnaire. Sleep will be assessed by sleep logs and actigraphy for sleep onset time, sleep latency, total sleep time, total wake time, number and length of awakenings, sleep efficiency, sleep fragmentation index and sleep mean activity score. Recovery measures will include: length of hospitalization, infection rate, body temperature, cortisol levels, cooperation with medical staff.

Study plan. The research will comprise of 5 consecutive steps. Step 1 will include the week prior to surgery and include sleep evaluation to all participants by sleep log and actigraphy. Step 2 is the night prior to surgery and will include sleep log and actigraphy. 30 children will receive melatonin (Circadin) 2mg, 30 children will receive placebo and 30 children will constitute the control group. Step 3 will be conducted during anesthesia and surgery where stress variables and need for anesthesia will be recorded. Step 4 will take place during post-operative hospitalization and will include actigraphy and sleep logs. Step 5 will take place at home two weeks after discharge and will include actigraphy and sleep logs.

DETAILED DESCRIPTION:
Data for each participant will be collected from the medical records and will include: demographic data, gender, and clinical background. Underlying sleep disorders will be screened by an accepted and validated sleep questionnaire [28] (appendix A) The study will consist of 5 sequential and continual steps: step 1 - the week prior to admission to the hospital; step 2 - the night before surgery; step 3 - anesthesia and surgery; step 4 - the post operative hospital stay; step 5 - home, 2 weeks after discharge.

Step 1: all 90 patients will undergo sleep evaluation by actigraphy and a sleep log (appendix B), for 7 days prior to surgery in their usual sleep environment at home.

Step 2: the patients will be divided into 3 study groups in a double-blind, placebo-controlled randomization:

1. Thirty children will receive melatonin (Circadin) 2 mg, one hour before bedtime and will consist of study group A.
2. Thirty age, gender and disease matched controls will receive placebo and will consist of placebo group A.
3. Thirty age, gender and disease matched children will not receive anything (control group).

Actigraphy and completion of sleep questionnaire will be also performed in hospital in the night prior to surgery.

Step 3: stress assessment during anesthesia and surgery will be assessed by the following variables that are routinely monitored and recorded during surgery by the MDsoft computerized system: heart rate, blood pressure, end-tidal CO2, amount of anesthetic agents, opiate consumption.

Step 4: actigraphy and completion of sleep questionnaire will be performed in each night of the post-surgery hospital stay period and up to 1 week post-surgery.

Step 5: two weeks after discharge, an additional follow-up sleep log and actigraphy will be performed for 5 consecutive nights.

Practically, children will be recruited in triplicates so that each triple will consist of the same gender, age and type of surgery. By randomization they will be assigned to one of each of the study groups.

Post operatively, each pair of patients of study group A and the placebo group A (not including control group) will be randomly re-divided into two new groups: study group B - children who will receive melatonin every night and control group B who will receive placebo every night one hour before bedtime for the rest of the hospitalization.

Sleep evaluation:

Sleep will be evaluated by sleep log which is a diary of sleep variables completed by parents after each night (appendix B) and by actigraphy.

Actigraphy An actigraph is a watch-like device that is placed on the wrist. It is a noninvasive continuous ambulatory measure used to objectively evaluate sleep. The use of actigraphy for both clinical and research purposes is well established. Actigraphy is a reliable and valid tool for detecting disturbed sleep and a useful technique for the evaluation of insomnia and circadian rhythm disorders [10]. It is an accepted and common technique in children [29] and is routinely used in our pediatric sleep clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age: 4-18 years scheduled for elective surgery in the general pediatric surgery, pediatric orthopedics, pediatric urology and the pediatric plastic departments

Exclusion Criteria:

* An underlying known sleep disorder such as delayed sleep phase syndrome, sleep-disordered breathing and insomnia
* An underlying medical condition that may directly affect sleep (state of decreased consciousness, brain surgery)
* Taking medications that may affect sleep
* Impairment of renal or liver functions
* Autoimmune diseases
* Known galactose intolerance, lactase deficiency, glucose-galactose malabsorption

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency | 1. Night before surgery, 2. Nights in hospital after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel